CLINICAL TRIAL: NCT04989777
Title: The Effect of IABP in the Early Stage of Acute Myocardial Infarction With Cardiogenic Shock (SCAI-B): a Multicenter, Prospective, Randomized Controlled Study
Brief Title: IABP In AMI Patients With SCAI-B Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 68752
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Myocardial Infarction, Acute; Cardiogenic Shock
Keywords: IABP; Acute myocardial infarction; cardiogenic shock; SCAI-B
MeSH Terms: conditions — Myocardial Infarction; Shock, Cardiogenic | interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients with AMI and shock stage B were received Standardized treatment
- IABP group (Experimental): Patients with AMI and shock stage B were received Standardized treatment and IABP treatment
  Interventions: Device: IABP (Intra-aortic balloon pump ) implantation

INTERVENTIONS:
Device: IABP (Intra-aortic balloon pump ) implantation — Eligible AMI patients in SCAI-B stage will receive IABP implantation from the femoral artery
  Arms: IABP group

SUMMARY:
Acute myocardial infarction (AMI) is the most common cause of cardiogenic shock (CS), and CS is the most common cause of death in patients with AMI. Percutaneous mechanical circulation is one of the most important techniques in the treatment of AMICS. Intra-aortic balloon pump (IABP) is the most commonly used mechanical circulatory assist device in clinic. However, the existing clinical evidence shows that IABP can not improve the clinical outcome of patients with AMICS. As for impella and extracorporeal membrane oxygenation (ECMO) system, there was still no difference in overall mortality compared with IABP in AMICS.

Until now, IABP-shock II study is the largest randomized controlled study so far. However, this study has limitations. In a recent retrospective study, the project team investigated the use of IABP and the outcomes of more than 300 AMI cases in three provincial capitals of Northeast China in 2016. It was found that the 28 day survival rate of patients in the early use of IABP group was significantly higher than that in the late use group. The investigators speculate that IABP may significantly improve the clinical outcomes of patients with AMICS if it can be used in the earlier stage of CS (stage B).

This multicenter, prospective, randomized controlled study will involve 512 participants in about 15 centers. Patients diagnosed with AMI (including STEMI and NSTEMI) complicated with shock stage B (SCAI definition criteria) received early revascularization (PCI or CABG) and standardized drug treatment according to the current guidelines before meeting the study inclusion criteria. After reviewing the inclusion criteria, participants were randomized to two groups (IABP group and control group) in a ratio of 1:1.

The investigators speculated that IABP could significantly improve the clinical outcomes of patients with AMICS if it could be used in the earlier stage of CS (stage B). At present, there is no clinical study on the use of IABP in AMICS (stage B). It is worth carrying out the corresponding clinical research, in order to study the real role of IABP in patients with AMICS and explore the treatment strategy of AMICS in line with China's national conditions.

DETAILED DESCRIPTION:
(A).Background AMICS is the most common cause of death in patients with coronary heart disease. Even with modern treatment, including early reperfusion combined with mechanical assistive devices, the 30-day mortality of AMICS is still close to 50%. At present, mechanical assistive devices mainly include IABP, ECMO, and impalla.

As far as China's national conditions are concerned, IABP is still the most easily available mechanical assistive device for clinical operation and management. IABP can reduce cardiac afterload, decrease myocardial oxygen consumption and increase cardiac output in patients with AMICS, which is helpful to protect the myocardium and improve end-organ perfusion. In previous registration studies or retrospective analyses on IABP, the mortality of CS patients using IABP was significantly lower than that of the control group. Therefore, the use of IABP in patients with AMICS are class I recommendations in the early (before 2012) American and European guidelines. Until 2012, the results of IABP-SHOCK II study were released, the effect of IABP on patients with AMICS began to be questioned. IABP-SHOCK II study is the largest randomized controlled study so far. Compared with traditional treatment, IABP did not improve AMICS mortality in 30 days, 1 year, and 6 years. Subsequently, European guidelines did not recommend routine use of IABP (level III recommendation) in AMICS, while American guidelines changed from level I recommendation to level IIb recommendation . However, the IABP-SHOCK II study has some limitations: (1) the severity of CS in the patients included in this study varies greatly; (2) IABP was used relatively late (most patients received IABP treatment after revascularization and severe tissue hypoperfusion).

CS patients are a heterogeneous population, and the prognosis may vary greatly with the severity of shock. In order to guide treatment and predict clinical outcomes more accurately, the consensus statement of clinical experts on classification of cardiogenic shock SCAI was issued at the 42nd Annual Meeting of angiocardiography and intervention (SCAI) in 2019, which divided CS into five stages: a (risk stage), B (initial stage), C (typical stage), D (deterioration stage) and E (end stage). In the IABP-SHOCK II study, the inclusion criteria of CS patients were (1) systolic blood pressure < 90mmHg for more than 30min or the need for catecholamine drugs to maintain systolic blood pressure > 90mmHg with signs of pulmonary congestion; (2) The symptoms of organ hypoperfusion (at least in accordance with the following 1 item): (a) change of mental state; (b) The limbs and skin are cold and wet; (c) The decrease of urine volume was less than 30ml / h; (d) Lactic acid > 2.0mmol/l. Therefore, patients with CS of stage C (typical stage) or more severity were included in IABP-SHOCK II study. According to the "Chinese expert consensus on diagnosis and treatment of cardiogenic shock (2018)", it is emphasized that IABP should be implanted as soon as possible and maintained for enough time in patients with AMICS. In addition, in a recent retrospective study, the project team investigated the use of IABP and the outcomes of more than 300 AMI cases in three provincial capitals of Northeast China in 2016. It was found that the 28-day survival rate of patients in the early use of IABP group was significantly higher than that in the late use group.

The investigators speculated that IABP could significantly improve the clinical outcomes of patients with AMICS if it could be used in the earlier stage of CS (stage B). At present, there is no clinical study on the use of IABP in AMICS (stage B). It is worth carrying out the corresponding clinical research, in order to study the real role of IABP in patients with AMICS and explore the treatment strategy of AMICS in line with China's national conditions.

(B).Preliminary Data The clinical data of all patients receiving IABP treatment in 8 top three hospitals in three provincial capitals of Northeast China. The reasons for receiving IABP treatment, the duration of treatment and the clinical outcomes of patients were recorded. At the same time, the high-risk PCI patients were analyzed according to early IABP implantation (before PCI or at the same time) and late implantation (after PCI).

Only one of the eight hospitals is a heart center with more than 2000 cases of operation and more than 200 cases of IABP implantation. The 28 day survival rate of patients with IABP implantation is 87.9%, which is significantly higher than that of other hospitals. IABP is widely used in high-risk PCI patients (77.5% of left main coronary artery disease, 13.9% of multi vessel disease), patients with acute myocardial infarction ventricular septal perforation and unable to carry out revascularization, and patients with severe myocarditis. IABP treatment time is 12-186 hours, 28 day survival rate is 78.2%. Especially, the survival rate of early IABP implantation was significantly higher than that of late group (89% vs. 63%, P < 0.05) in high risk AMI with left main and multi-vessel lesions

(C). Research Design and Methodology This multicenter, prospective, randomized controlled study will involve 512 participants in about 15 centers. Patients diagnosed with AMI (including STEMI and NSTEMI) complicated with shock stage B (SCAI definition criteria) received early revascularization (PCI or CABG) and standardized drug treatment according to the current guidelines before meeting the study inclusion criteria. After reviewing the inclusion criteria, participants were randomized to two groups (IABP group and control group) in a ratio of 1:1.

1. Inclusion criteria (1) Patients aged 18-85 years with AMI (STEMI or NSTEMI) and shock stage B (SCAI definition criteria); (2) Plan to implement revascularization (PCI or CABG) (3) Hypotension: SBP < 90mmHg or map < 60mmhg or decrease > 30mmhg from baseline, more than 30min under the condition of sufficient blood volume; (4) No signs of hypoperfusion (if one of the following conditions is met): :1) Good mental state; 2) The extremities were warm without cold and wet; 3) Lactic acid ≤ 2 mm; 4) Normal renal function or mild renal impairment (creatinine increase less than one time or GFR decrease ≤ 50%.
2. Exclusion criteria (1) Age > 85; (2) CPR > 30 min; (3) Stage C-E in SCAI shock definition criteria; (4) Acute pulmonary embolism; (5) Mechanical complications, such as ventricular septal perforation, acute mitral regurgitation; (6) Non drug induced severe central nervous system dysfunction; (7) Other causes of shock, such as septic shock, hemorrhagic shock, ketoacidosis; (8) Aortic insufficiency above grade II; (9) Difficulty in IABP implantation due to severe peripheral vascular disease; (10) Combined with other serious diseases and life expectancy < 12 months; (11) Refusal to sign informed consent
3. Study endpoint

(1) Primary endpoint: 30 day all-cause death (2) Secondary endpoint

1. Key secondary endpoints: all cause death, cardiac death, readmission of heart failure, NYHA I / II ratio of cardiac function, KCQQ score.
2. Other secondary end points: ① Monitoring treatment parameters: the proportion of shock progressing to SCAI stage C / D / E, the time required for hemodynamic stability, the dosage and type of vasoactive drugs, the length of stay in CCU unit, and the use rate of more advanced cardiac assistive devices (ECMO and impalar). ② Myocardial perfusion and microcirculation flow score.

(3) Primary safety end point: Gusto defined massive or life-threatening bleeding, disabling stroke, peripheral vascular complications requiring surgical or interventional treatment.

4. Statistical analysis

1. Sample size estimation According to the results of previous studies on SCAI shock, the retrospective statistical results of the three northeastern provinces in the early stage of IABP and the recommendations of the expert group, it is estimated that the event rate of the control group is 34%, and that of the IABP group is 22%. In order to detect the relative risk of 35% reduction in bilateral α According to the statistical power calculation of 5% and 80%, and considering the shedding rate of 10%, 256 patients / group (a total of 512 patients) were calculated.
2. Effectiveness and safety analysis The measurement data and counting data passed t test, chi square test or Fisher test. Survival analysis was used to describe the primary and secondary endpoints. Log rank sum test was used for comparison between the study groups. Cox proportional hazards regression model was used to estimate the risk ratio of each endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-85 years with AMI (STEMI or NSTEMI) and shock stage B (SCAI definition criteria)
2. Plan to implement revascularization (PCI or CABG)
3. Hypotension: SBP < 90mmHg or map < 60mmhg or decrease > 30mmhg from baseline, more than 30min under the condition of sufficient blood volume; (4) No signs of hypoperfusion (if one of the following conditions is met):1) Good mental state; 2) The extremities were warm without cold and wet; 3) Lactic acid ≤ 2 mm; 4) Normal renal function or mild renal impairment (creatinine increase less than one time or GFR decrease ≤ 50%.

Exclusion Criteria:

1. Age > 85
2. CPR > 30 min
3. Stage C-E in SCAI shock definition criteria
4. Acute pulmonary embolism
5. Mechanical complications, such as ventricular septal perforation, acute mitral regurgitation
6. Non-drug induced severe central nervous system dysfunction
7. Other causes of shock, such as septic shock, hemorrhagic shock, ketoacidosis
8. Aortic insufficiency above grade II
9. Difficulty in IABP implantation due to severe peripheral vascular disease
10. Combined with other serious diseases and life expectancy < 12 months
11. Refusal to sign the informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Event | In-hospital 30-day
  All-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Cheng, Study Director — Renmin Hospital of Wuhan University
Locations (1):
- Renmin hospital of Wuhan university, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goldberg RJ, Spencer FA, Gore JM, Lessard D, Yarzebski J. Thirty-year trends (1975 to 2005) in the magnitude of, management of, and hospital death rates associated with cardiogenic shock in patients with acute myocardial infarction: a population-based perspective. Circulation. 2009 Mar 10;119(9):1211-9. doi: 10.1161/CIRCULATIONAHA.108.814947. Epub 2009 Feb 23. PMID 19237658
- [Result] Barron HV, Every NR, Parsons LS, Angeja B, Goldberg RJ, Gore JM, Chou TM; Investigators in the National Registry of Myocardial Infarction 2. The use of intra-aortic balloon counterpulsation in patients with cardiogenic shock complicating acute myocardial infarction: data from the National Registry of Myocardial Infarction 2. Am Heart J. 2001 Jun;141(6):933-9. doi: 10.1067/mhj.2001.115295. PMID 11376306
- [Result] Antman EM, Anbe DT, Armstrong PW, Bates ER, Green LA, Hand M, Hochman JS, Krumholz HM, Kushner FG, Lamas GA, Mullany CJ, Ornato JP, Pearle DL, Sloan MA, Smith SC Jr, Alpert JS, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Gregoratos G, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 1999 Guidelines for the Management of Patients With Acute Myocardial Infarction). ACC/AHA guidelines for the management of patients with ST-elevation myocardial infarction--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 1999 Guidelines for the Management of Patients With Acute Myocardial Infarction). Circulation. 2004 Aug 3;110(5):588-636. doi: 10.1161/01.CIR.0000134791.68010.FA. No abstract available. PMID 15289388
- [Result] Van de Werf F, Bax J, Betriu A, Blomstrom-Lundqvist C, Crea F, Falk V, Filippatos G, Fox K, Huber K, Kastrati A, Rosengren A, Steg PG, Tubaro M, Verheugt F, Weidinger F, Weis M; ESC Committee for Practice Guidelines (CPG). Management of acute myocardial infarction in patients presenting with persistent ST-segment elevation: the Task Force on the Management of ST-Segment Elevation Acute Myocardial Infarction of the European Society of Cardiology. Eur Heart J. 2008 Dec;29(23):2909-45. doi: 10.1093/eurheartj/ehn416. Epub 2008 Nov 12. No abstract available. PMID 19004841
- [Result] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, de Waha A, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Lauer B, Bohm M, Ebelt H, Schneider S, Werdan K, Schuler G; Intraaortic Balloon Pump in cardiogenic shock II (IABP-SHOCK II) trial investigators. Intra-aortic balloon counterpulsation in acute myocardial infarction complicated by cardiogenic shock (IABP-SHOCK II): final 12 month results of a randomised, open-label trial. Lancet. 2013 Nov 16;382(9905):1638-45. doi: 10.1016/S0140-6736(13)61783-3. Epub 2013 Sep 3. PMID 24011548
- [Result] Thiele H, Zeymer U, Thelemann N, Neumann FJ, Hausleiter J, Abdel-Wahab M, Meyer-Saraei R, Fuernau G, Eitel I, Hambrecht R, Bohm M, Werdan K, Felix SB, Hennersdorf M, Schneider S, Ouarrak T, Desch S, de Waha-Thiele S; IABP-SHOCK II Trial (Intraaortic Balloon Pump in Cardiogenic Shock II) Investigators; IABP-SHOCK II Investigators. Intraaortic Balloon Pump in Cardiogenic Shock Complicating Acute Myocardial Infarction: Long-Term 6-Year Outcome of the Randomized IABP-SHOCK II Trial. Circulation. 2019 Jan 15;139(3):395-403. doi: 10.1161/CIRCULATIONAHA.118.038201. Epub 2018 Nov 11. PMID 30586721
- [Result] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Ting HH, O'Gara PT, Kushner FG, Ascheim DD, Brindis RG, Casey DE Jr, Chung MK, de Lemos JA, Diercks DB, Fang JC, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2015 ACC/AHA/SCAI Focused Update on Primary Percutaneous Coronary Intervention for Patients With ST-Elevation Myocardial Infarction: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention and the 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction. J Am Coll Cardiol. 2016 Mar 15;67(10):1235-1250. doi: 10.1016/j.jacc.2015.10.005. Epub 2015 Oct 21. No abstract available. PMID 26498666
- [Result] Henry TD, Tomey MI, Tamis-Holland JE, Thiele H, Rao SV, Menon V, Klein DG, Naka Y, Pina IL, Kapur NK, Dangas GD; American Heart Association Interventional Cardiovascular Care Committee of the Council on Clinical Cardiology; Council on Arteriosclerosis, Thrombosis and Vascular Biology; and Council on Cardiovascular and Stroke Nursing. Invasive Management of Acute Myocardial Infarction Complicated by Cardiogenic Shock: A Scientific Statement From the American Heart Association. Circulation. 2021 Apr 13;143(15):e815-e829. doi: 10.1161/CIR.0000000000000959. Epub 2021 Mar 4. PMID 33657830
- [Result] Baran DA, Grines CL, Bailey S, Burkhoff D, Hall SA, Henry TD, Hollenberg SM, Kapur NK, O'Neill W, Ornato JP, Stelling K, Thiele H, van Diepen S, Naidu SS. SCAI clinical expert consensus statement on the classification of cardiogenic shock: This document was endorsed by the American College of Cardiology (ACC), the American Heart Association (AHA), the Society of Critical Care Medicine (SCCM), and the Society of Thoracic Surgeons (STS) in April 2019. Catheter Cardiovasc Interv. 2019 Jul 1;94(1):29-37. doi: 10.1002/ccd.28329. Epub 2019 May 19. PMID 31104355
- [Result] Subspecialty Group of Acute and Intensive Cardiac Care of Chinese Society of Cardiology; Editorial Board of Chinese Journal of Cardiology. [Chinese experts consensus on the diagnosis and treatment of cardiogenic shock(2018)]. Zhonghua Xin Xue Guan Bing Za Zhi. 2019 Apr 24;47(4):265-277. doi: 10.3760/cma.j.issn.0253-3758.2019.04.003. Chinese. PMID 31060185